CLINICAL TRIAL: NCT00886678
Title: A Phase II Study of Pemetrexed Plus Carboplatin Combined With Radiation in Patients With Inoperable Locally Advanced Non-small Cell Lung Cancer
Brief Title: A Study of Pemetrexed Plus Carboplatin Combined With Radiation in Patients With Inoperable Locally Advanced Non-small Cell Lung Cancer (LA-NSCLC) (RT0801)
Acronym: NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Ma Shenglin, Xu Yaping, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH01
Record Dates: First submitted 2009-03-31; First posted 2009-04-23 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2010-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; pemetrexed; radiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): patients receiving pemetrexed, carboplatin and radiation therapy.
  Interventions: Drug: pemetrexed; Drug: carboplatin; Radiation: thoracic radiation

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2, IV, q 21 days x 2 cycles
Drug: carboplatin — AUC=5,IV,q 21 days x 2 cycles
Radiation: thoracic radiation — 66 Gy over 33 fractions

SUMMARY:
Patients with inoperable Non-Small-Cell Lung Cancer will receive thoracic radiation therapy 66 Gy over 33 fractions,and concurrent with 2 cycles of chemotherapy with pemetrexed (500 mg/m2,d1,repeated every 3 weeks)and carboplatin (AUC=5,d1,repeated every 3 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small cell lung cancer (non-squamous cell carcinoma)
* Presence of measurable disease by RECIST
* Inoperable stage IIIA or IIIB
* ECOG performance status 0-1
* No prior chemotherapy, radiation therapy to chest, immunotherapy, or biologic therapy
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital.

Exclusion Criteria:

* Carcinoid tumor, small cell carcinoma of lung
* Patients with any distant metastasis
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix Any other morbidity or situation with contraindication for chemotherapy (e.g. active infection, myocardial infarction preceding 6 months, symptomatic heart disease including unstable angina, congestive heart failure or uncontrolled arrhythmias, immunosuppressive treatment)
* Pregnant or lactating women, women who has not taken test of pregnancy (within 14 days before the first administration) and pregnant women
* Women and men of childbearing potential who have no willing of employing adequate contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
tumor response rate | Tumor assessments after completion of chemoradiotherapy and every 2 months

SECONDARY OUTCOMES:
overall survival | baseline to date of death from any cause
time to progressive disease | baseline to measured progressive disease
the safety profile | every cycle
site of first failure in patients who develop progressive disease | baseline to measured progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Ma Sheng lin, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China